CLINICAL TRIAL: NCT01566981
Title: E-support for Healthcare Processes - DIABETES
Brief Title: E-health Care Process Support for Diabetes Type II Patients
Acronym: EHDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Collaborators: University of Ljubljana School of Medicine, Slovenia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EHDI
Record Dates: First submitted 2012-02-12; First posted 2012-03-30 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus Type II,
Keywords: Diabetes mellitus tip II; eHealth solution; Health Information Technology; quality of life; family medicine; satisfaction with e-health care; primary care
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Primary Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diabetes with ICT support (E-diabetes) (Experimental): The group of randomly selected patients with DM type II, who will get the software application and web- based support Intervention: Computerised support to the Diabetes type II patients
  Interventions: Procedure: Computerised support to the Diabetes type II patients
- Diabetes without support (No Intervention): The group of randomly selected patients with DM type II, without software application and web-based support.

INTERVENTIONS:
Procedure: Computerised support to the Diabetes type II patients — The randomly selected group of patients with diabetes type II will get software application and web based support to their usual healthcare process.
  Other Names: eDiabetes in Primary healthcare
  Arms: Diabetes with ICT support (E-diabetes)

SUMMARY:
The purpose of the study is to clinically evaluate a new approach to treatment of patients with diabetes mellitus type II by using specially developed mobile-internet software solution.

The effect of information and communication technologies (ICT) to improve the integrated care of people with diabetes will be identified, developed, introduced and clinically evaluated.

The investigators expect that usage of an e-Health application in health care of patients with diabetes mellitus type II could improve the following healthcare outcomes: results of the laboratory tests (with emphasis on HbA1C value), regular medication usage, blood pressure values, Body mass index (BMI) values, diet, regular exercise and quality of life.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is defined as a "group of common metabolic disorders that share the phenotype of hyperglycemia". It is generally agreed that in Caucasian populations the prevalence rate is between 2% and 6%. Prevalence rate of DM in SLovenia is about 5%. Type 2 DM accounts for 90% to 95% of all diabetes cases.

Results of many clinical studies demonstrated the great potential of information and communication technology (ICT) applications to improve health care of patients with chronic diseases including diabetes mellitus.

In this study an ICT mobile environment to improve the process of an integrated care of people with Diabetes mellitus will be identified, developed, introduced and clinically evaluated. The study will include 140 patients diagnosed with diabetes mellitus type II who are managed in primary care. The study will use and evaluation questionnaire that will cover issues regarding the patient quality of life.

Subjects with a blood pressure meter and a scale, will be able to enter the value of the systolic and diastolic blood pressure and the body weight.

Subjects will be motivated to regularly enter data about their blood pressure, body weight, dietary misconducts and to complete available questioners. In addition to this, users can enter values about their physical activity (type, duration, intensity).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, treated with non-pharmacological interventions or/and tablets (Non-Insulin-Dependent Diabetes Mellitus)
* Internet connection and personal computer /lap-top computer
* Mobile phone
* Sufficient level of Internet and e-mail usage - checked by short questionnaire
* Age >18 or <75 years

Exclusion Criteria:

* significant co-morbidity
* Type 1 diabetes
* Insulin-dependent type 2 diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Brodnik, PhD, Principal Investigator — University of Ljubljana, FRI and University of Primorska, DIST
Locations (2):
- Slovenia (2):
  - Department of family medicine in Ljubljana, Ljubljana
  - Department of Family medicine, Medical Faculty, Ljubljana

RESULTS

PARTICIPANT FLOW:
Groups:
- Diabetes With ICT Support (E-diabetes): The group of randomly selected patients with DM type II, who will get the software application and web- based support Intervention: Computerised support to the Diabetes type II patients
  Computerised support to the Diabetes type II patients: 58 randomly selected patients with diabetes type II got software application and web based support to their usual healthcare process.
  5 patients were lost to follow up, consequently 53 patients were included in final analysis
- Diabetes Without Support: 62 randomly selected patients with DM type II that were followed by using usual healthcare - without software application and web-based support.
  8 patients were lost to follow up, so 54 patients were included in final analysis.
Period: Overall Study
Arm/Group | Diabetes With ICT Support (E-diabetes) | Diabetes Without Support
Started | 58 | 62
Completed | 53 | 54
Not Completed | 5 | 8
Not completed — Lost to Follow-up | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Diabetes With ICT Support (E-diabetes): The group of randomly selected patients with Diabetes mellitus (DM) type II, who will get the software application and web- based support Intervention: Computerized support to the Diabetes type II patients
  Computerized support to the Diabetes type II patients: The randomly selected group of patients with diabetes type II will get software application and web based support to their usual healthcare process.
- Total: Total of all reporting groups
Arm/Group | Diabetes With ICT Support (E-diabetes) | Diabetes Without Support | Total
Number analyzed (Participants) | 58 | 62 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (10.5) | 54.7 (11.1) | 55.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 47
  Male | 36 | 37 | 73
Years of DM treatment [Mean (Standard Deviation); unit: years] | 5.1 (5.7) | 5.7 (4.8) | 5.5 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1C at 1 Year.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percentage of glycated haemoglobin
Groups:
- Diabetes Without Support: 62 randomly selected patients with DM type II that were followed by using usual healthcare - without software application and web-based support.
  8 patients were lost to follow and 54 patients were included in final analysis.
Arm/Group | Diabetes With ICT Support (E-diabetes) | Diabetes Without Support
Number analyzed (Participants) | 53 | 54
percentage of glycated haemoglobin | 0.6925 (1.4708) | 0.1707 (1.0617)
Statistical Analysis 1: Comparison: Diabetes With ICT Support (E-diabetes); Null hypothesis was that Information and Communication Technology (ICT) supported diabetes care could have significant impact on reduction of baseline glycated hemoglobin (EHbA1c) after 1 year follow-up. The sample in intervention group was normally distributed, so observed power (two-tailed hypothesis) was 0.45, for Cohen's d= 0.6 and alpha level =0.05; Test type: Superiority or Other; p = 0.005, t-test, 2 sided; without adjustments, df=39; Mean Difference (Final Values) = 0.6925, 95% CI 2-sided [0.2221 to 1.1629], Standard Deviation 1.4708

2. Secondary Outcome: Body Mass Index at 1 Year
Time Frame: one year
Measure: Mean (Standard Deviation); unit: Kg/m2
Arm/Group | Diabetes Without Support | Diabetes With ICT Support (E-diabetes)
Number analyzed (Participants) | 54 | 53
Kg/m2 | 31.76 (4.87) | 32.6 (5.14)

3. Secondary Outcome: Patients' Functional Health Status Via WONCA-COOP Questionnaire.
Description: WONCA COOP questionnaire measure seven core aspects of functional status, therefore this instrument consists of 7 five-point ordinal sub-scales. Each scale ranging from 1 ('no limitation at all') to 5 ('severely limited'); for 'change in health' score 1 means 'much better' and score 5'much worse'. Sub-scales are averaged to compute a total score.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diabetes With ICT Support (E-diabetes) | Diabetes Without Support
Number analyzed (Participants) | 53 | 54
units on a scale | 2.12 (0.66) | 1.89 (0.58)

4. Secondary Outcome: Change of Blood Lipid Level ( Low Density Cholesterol)
Time Frame: baseline and one year
Reporting Status: Not Posted

5. Secondary Outcome: Quality of Patients' Life Via WONCA-COOP Questionnaire.
Time Frame: baseline and one year
Reporting Status: Not Posted

6. Secondary Outcome: Change of Patients' Functional Health Status Via WONCA-COOP Questionnaire.
Time Frame: baseline and one year
Reporting Status: Not Posted, anticipated posting 2013-11

7. Secondary Outcome: Change of Blood Lipid Level ( Low Density Cholesterol)
Time Frame: baseline and six months
Reporting Status: Not Posted

8. Secondary Outcome: Change of the Following Parameter : HbA1C
Time Frame: baseline and six months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 15 months
Groups:
- Diabetes With ICT Support (E-diabetes): The group of randomly selected patients with DM type II, who will get the software application and web- based support Intervention: Computerised support to the Diabetes type II patients
  Computerised support to the Diabetes type II patients: 58 randomly selected patients with diabetes type II got software application and web based support to their usual healthcare process.
  5 patients were lost to follow up and 13 patients missed final consultation, consequently 53 patients were included in final analysis
- Diabetes Without Support: 62 randomly selected patients with DM type II that were followed by using usual healthcare - without software application and web-based support.
  8 patients were lost to follow up and 12 patients missed final consultation. 54 patients were included in final analysis.
Arm/Group | Diabetes With ICT Support (E-diabetes) | Diabetes Without Support
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/62
Other Adverse Events (participants affected / at risk) | 0/58 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No